CLINICAL TRIAL: NCT04444752
Title: A Randomized, Double-Blind, Placebo-Controlled Multi-Centered Study of the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of CBP-201 in Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Assess the Efficacy and Safety of CBP-201 in Adult Subjects With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-201-WW001
Record Dates: First submitted 2020-06-15; First posted 2020-06-24 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CBP-201 Dose 1 (Experimental): CBP-201 Dose 1 subcutaneous (SC) injection
  Interventions: Drug: CBP-201
- CBP-201 Dose 2 (Experimental): CBP-201 Dose 2 subcutaneous (SC) injection
  Interventions: Drug: CBP-201
- CBP-201 Dose 3 (Experimental): CBP-201 Dose 3 subcutaneous (SC) injection
  Interventions: Drug: CBP-201
- placebo (Placebo Comparator): subcutaneous (SC) injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CBP-201 — CBP-201 subcutaneous(SC) injection.
  Arms: CBP-201 Dose 1; CBP-201 Dose 2; CBP-201 Dose 3
Drug: placebo — subcutaneous(SC) injection
  Arms: placebo

SUMMARY:
This study will evaluate the efficacy, safety, pharmacokinetics and pharmacodynamics of CBP-201 in adult subjects with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose regimen finding study to assess the efficacy, safety, and steady-state PK profile of CBP-201 administered to eligible adult subjects with moderate to severe atopic dermatitis compared to placebo. CBP-201 is administered as a subcutaneous (SC) injection. The study is divided into a treatment period of 16 weeks and a follow-up period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be an adult ≥18 and ≤ 75 years of age at the screening visit (Screening) with atopic dermatitis according to American Academy of Dermatology Consensus Criteria, (Eichenfield 2014)
2. Present for at least 1 year prior to the baseline visit (Baseline) with an inadequate response, in the judgement of the Investigator, to AD treatment with a topical regimen of corticosteroids, phosphodiesterase inhibitors or calcineurin inhibitors, or for whom topical treatments are otherwise medically inadvisable (eg, because of important side effect or safety risks)
3. Investigator Global Assessment (IGA) score ≥ 3 at Screening and Baseline.
4. Eczema Area and Severity Index (EASI) score ≥ 16 at Screening and Baseline
5. Body Surface Area (BSA) for total AD involvement ≥ 10% at Screening and Baseline
6. Able and willing to apply a stable dose of a bland emollient twice a day to affected areas for at least 7 days before Baseline and to continue for the duration of the study
7. Females of child-bearing potential (FCBP) and males who have not undergone a vasectomy must abstain from heterosexual activities or agree to use effective contraception throughout the entire study period.

Exclusion Criteria:

1. Have any of the following laboratory abnormalities at Screening:

   1. Hemoglobin ≤ 90% of the lower limit of normal range (LLN)
   2. White blood cell (WBC) below the LLN
   3. Neutrophil count below the LLN
   4. Platelet count below the LLN
2. Have undergone treatment with any of the following:

   1. Topical agents such as corticosteroids, phosphodiesterase (PDE) inhibitors, Janus kinase (JAK) inhibitors, tacrolimus or pimecrolimus within 1 week prior to Baseline. Note that low to medium potency topical corticosteroids (TCS) are permitted after randomization to treat AD flares
   2. Prior treatment with dupilumab or any antibody against IL-4Rα or IL-13
   3. Systemic treatment for AD or other condition with steroids or other immunosuppressive/immunomodulating substances, e.g., cyclosporine, mycophenolate-mofetil, azathioprine, methotrexate or oral Janus kinase (JAK) inhibitors within 4 weeks prior to Baseline. Use of steroid inhalers and nasal corticosteroids is allowed.
   4. Cell depleting agents, e.g. rituximab, within 6 months of Baseline or treatment with other biologics within 5 half-lives (if known) or 3 months prior to baseline visit, whichever is longer
   5. Phototherapy (narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + ultraviolet A [PUVA]), tanning beds, or any other light emitting device (LED), within 4 weeks of Baseline
   6. ≥ 2 bleach baths within 2 weeks of Baseline
   7. Prescription emollient to treat AD (e.g. Atopiclair®, MimyX®, Epicerum®, etc.) within 2 weeks of Baseline
   8. Any investigational drug within 30 days or within 5 half-lives, whichever is longer, before Baseline.
   9. Live (attenuated) vaccine within 8 weeks of Baseline.
   10. Treatment with systemic traditional Chinese medicine (TCM) or herbal medications within 4 weeks before Baseline or treatment with topical TCM or herbal medications within 1 week before Baseline visit
3. Have any of the following:

   1. Infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks before Baseline, or superficial skin infection, such as impetigo, within 2 weeks before the Baseline (subjects may be rescreened after the infection has resolved)
   2. A history of parasitic infection (e.g. helminth), within 6 months of Baseline
   3. Per investigator judgement, known or suspected history of immunosuppression within 6 months of Baseline, including a history of invasive opportunistic infections, such as aspergillosis, coccidioidomycosis, histoplasmosis, human immunodeficiency virus (HIV), listeriosis, pneumocystosis, or tuberculosis, despite infection resolution; or unusually frequent, recurrent or prolonged infections.
   4. Any history of vernal keratoconjunctivitis (VKC) and atopic keratoconjunctivitis (AKC)
   5. A history of malignancy with the following exceptions: completely treated carcinoma in situ of cervix or non-metastatic squamous or basal cell carcinoma of the skin
   6. Positive results at Screening for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibody with positive HCV RNA polymerase chain reaction; positive HIV serology at screening
   7. An allergy to L-histidine, trehalose or Tween (polysorbate) 80
4. Women must not be pregnant, planning to become pregnant or breast-feed during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzhou Connect, Study Director — Connect Biopharm LLC
Locations (59):
- United States (38):
  - Connect Investigative Site 310, Glendale, Arizona
  - Connect Investigative Site 338, Phoenix, Arizona
  - Connect Investigative Site 316, Tempe, Arizona
  - Connect Investigative Site 305, Little Rock, Arkansas
  - Connect Investigative Site 327, Canoga Park, California
  - Connect Investigative Site 324, Encinitas, California
  - Connect Investigative Site 301, Fremont, California
  - Connect Investigative Site 312, Huntington Beach, California
  - Connect Investigative Site 329, Mission Viejo, California
  - Connect Investigative Site 322, San Diego, California
  - Connect Investigative Site 323, San Luis Obispo, California
  - Connect Investigative Site 317, Santa Ana, California
  - Connect Investigative Site 318, Sherman Oaks, California
  - Connect Investigative Site 325, Thousand Oaks, California
  - Connect Investigative Site 332, Coral Gables, Florida
  - Connect Investigative Site 320, Hialeah, Florida
  - Connect Investigative Site 306, Hollywood, Florida
  - Connect Investigative Site 308, Jacksonville, Florida
  - Connect Investigative Site 314, Maitland, Florida
  - Connect Investigative Site 331, Miami, Florida
  - Connect Investigative Site 337, Miami, Florida
  - Connect Investigative Site 321, Miami, Florida
  - Connect Investigative Site 304, Orlando, Florida
  - Connect Investigative Site 340, Weston, Florida
  - Connect Investigative Site 333, Chicago, Illinois
  - Connect Investigative Site 303, Chicago, Illinois
  - Connect Investigative Site 307, New Albany, Indiana
  - Connect Investigative Site 313, West Lafayette, Indiana
  - Connect Investigative Site 311, Louisville, Kentucky
  - Connect Investigative Site 319, Hunt Valley, Maryland
  - Connect Investigative Site 335, Saint Joseph, Missouri
  - Connect Investigative Site 315, St Louis, Missouri
  - Connect Investigative Site 336, Las Vegas, Nevada
  - Connect Investigative Site 326, Albuquerque, New Mexico
  - Connect Investigative Site 330, Cincinnati, Ohio
  - Connect Investigative Site 328, Rapid City, South Dakota
  - Connect Investigative Site 309, Memphis, Tennessee
  - Connect Investigative Site 334, Houston, Texas
- Australia (8):
  - Connect Investigative Site 111, Canberra, Australian Capital Territory
  - Connect Investigative Site 104, Darlinghurst, New South Wales
  - Connect Investigative Site 108, Kanwal, New South Wales
  - Connect Investigative Site 105, Sydney, New South Wales
  - Connect Investigative Site 101, Brisbane, Queensland
  - Connect Investigative Site 102, Melbourne, Victoria
  - Connect Investigative Site 106, Fremantle, Western Australia
  - Connect Investigative Site 103, Perth, Western Australia
- China (9):
  - Connect Investigative Site 408, Beijing, Beijing Municipality
  - Connect Investigative Site 404, Beijing, Beijing Municipality
  - Connect Investigative Site 405, Wuxi, Jiangsu
  - Connect Investigative Site 409, Zhenjiang, Jiangsu
  - Connect Investigative Site 402, Jinan, Shandong
  - Connect Investigative Site 401, Shanghai, Shanghai Municipality
  - Connect Investigative Site 406, Shanghai, Shanghai Municipality
  - Connect Investigative Site 410, Tianjin, Tianjin Municipality
  - Connect Investigative Site 403, Hangzhou, Zhejiang
- New Zealand (4):
  - Connect Investigative Site 204, Tauranga, Bay of Plenty
  - Connect Investigative Site 202, Havelock North, Hawke's Bay Region
  - Connect Investigative Site 205, Waikanae, Kapiti Coast
  - Connect Investigative Site 203, Auckland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited based on physician referrral at academic and non-academic clinical centers between Jun 2020 and Sep 2021; 394 patients were screened. The first participant was randomized to treatment on 30 Jun 2020 and the last patient was randomized in April 2021. The last patient last visit was 22 Sept 2021.
Pre-assignment Details: After providing informed consent, patients were assessed for study eligibility within 45 days before the baseline visit. Of the 394 patients screeened, 226 patients met the eligibility criteria and were randomized to treatment.
Groups:
- CBP-201 150 Q2W: CBP-201 1800 mg, 600 mg Loading dose followed by 150 mg Q2W for 16 weeks
- CBP-201 300 Q2W: CBP-201 3000 mg, 600 mg Loading dose followed by 300 mg Q2W for 16 weeks
- CBP-201 300 Q4W: CBP-201 1800 mg, 600 mg Loading dose followed by 300 mg Q4W for 16 weeks alternating with 2 mLs matched volume placebo Q4W for 16 weeks
- Placebo: Placebo, 4 mLs matched loading dose volume follwed by 2 mls matched volume Q2W for 16 weeks
Period: Overall Study
Arm/Group | CBP-201 150 Q2W | CBP-201 300 Q2W | CBP-201 300 Q4W | Placebo
Started | 57 | 57 | 56 | 56
Completed | 46 | 45 | 50 | 40
Not Completed | 11 | 12 | 6 | 16
Not completed — Adverse Event | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 2 | 6 | 2 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 5 | 3 | 4
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Patient moving out of town | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBP-201 150 Q2W | CBP-201 300 Q2W | CBP-201 300 Q4W | Placebo | Total
Number analyzed (Participants) | 57 | 57 | 56 | 56 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 54 | 52 | 54 | 212
  >=65 years | 5 | 3 | 4 | 2 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (15.98) | 39.6 (14.79) | 41.7 (15.22) | 39.6 (14.79) | 40.1 (15.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 28 | 36 | 121
  Male | 27 | 30 | 28 | 20 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 24 | 27 | 24 | 92
  Not Hispanic or Latino | 40 | 33 | 29 | 32 | 134
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 17 | 9 | 12 | 14 | 52
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 1 | 3
  Black or African American | 8 | 7 | 10 | 6 | 31
  White | 30 | 38 | 32 | 32 | 132
  More than one race | 0 | 1 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  New Zealand | 5 | 3 | 5 | 6 | 19
  United States | 40 | 47 | 41 | 44 | 172
  China | 11 | 6 | 9 | 6 | 32
  Australia | 1 | 1 | 1 | 0 | 3
EASI Score [Mean (Standard Deviation); unit: units on a scale] — Eczema Area Severity Index Score
  units on a scale | 24.61 (10.471) | 27.57 (11.776) | 23.08 (8.218) | 25.16 (9.021) | 25.11 (10.042)
IGA Score [Count of Participants; unit: Participants]
  IGA 3 = Moderate disease | 43 | 34 | 40 | 39 | 156
  IGA 4 = Severe disease | 14 | 23 | 16 | 17 | 70
BSA [Mean (Standard Deviation); unit: percentage] — Body Surface Area affected by AD in %
  percentage | 39.86 (19.145) | 43.11 (20.738) | 37.34 (19.479) | 37.71 (18.341) | 39.52 (19.456)

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in EASI Score From Baseline to Week 16
Description: EASI=Eczema Area Severity Index is a validated physician score for signs of atopic dermatitis. EASI can range from 0 to 72. An EASI score of 0 indicates clear/no eczema, 0.1 to 1.0 almost clear, 1.1 to 7 mild disease, 7.1 to 21 moderate disease, 21.1 to 50 severe disease, and 51-72 indicates very severe disease. EASI Sub-scale ranges are as follows: Head/neck can range from 0-7.2, Trunk 0-14.4, Upper Extremities 0-21.6, Lower Extremities can range from 0-28.8. To calculate EASI, % involvement is first assessed by body region with an Area involvement Score of 0-6 for each region: 0=0%, 1=1-9%, 2=10-29%, 3=30-39%, 4=50-69%, 5=70-89%, 6=90-100% involvement. Then 4 attributes (Erythema, Edema/Papulation, Excoriation, and Lichenification) are scored for severity (0= none, 1=mild, 2=moderate, 3=severe). A multiplier is applied head/neck=0.1, trunk=0.2, upper extremities= 0.3, lower extremities=0.4. The total EASI score is the sum of 4 regional sub-scores.
Time Frame: Reduction from baseline to 16 weeks
Population: All efficacy analyses were carried out using the FAS (all randomized subjects who received at least part of an SC dose of study drug based on planned treatment assignment (ie, "as randomized").
Measure: Least Squares Mean (Standard Error); unit: percent reduction from Baseline
Arm/Group | CBP-201 150 Q2W | CBP-201 300 Q2W | CBP-201 300 Q4W | Placebo
Number analyzed (Participants) | 57 | 57 | 56 | 56
percent reduction from Baseline | 57.56 (4.610) | 63.03 (4.961) | 63.50 (4.661) | 39.67 (4.638)
Statistical Analysis 1: Comparison: CBP-201 300 Q2W vs Placebo; The primary efficacy analysis includes comparison of percentage reduction in EASI from baseline to Week 16 for CBP-201 300 mg Q2W regimen vs placebo. The sample size of the study was determined based on power calculations for the primary endpoint in patients receiving CBP-201 300 mg Q2W. Null hypothesis: CBP-201 300 Q2W is not superior to placebo in terms of percent reduction in EASI Score from Baseline to Week 16; Test type: Superiority — Pairwise comparisons for each CBP-201 group vs placebo were performed and a serial gate-keeping procedure was used for multiplicity adjustment. Each CBP-201 group was compared to placebo group in order from highest dose (300 mg Q2W) to the lowest dose frequency (300 mg Q4W), until statistical signficance at p=0.05 level was not achieved; p = 0.0007, ANCOVA — Adjusted for multiplicity using a serial gatekeeping procedure at the 5% in descending order: 1. 300 mg dose Q2W 2. 150 mg dose Q2W 3. 300 mg dose Q4W vs placebo; The data were analyzed using an ANCOVA model adjusted for treatment, baseline vIGA (moderate, severe), and baseline EASI; Mean Difference (Final Values) = 23.36, Standard Error of Mean 6.794
Statistical Analysis 2: Comparison: CBP-201 150 Q2W vs Placebo; The sample size of the study was determined based on power calculations for the primary endpoint in patients receiving CBP-201 300 mg Q2W. Null hypothesis: CBP-201 150 Q2W is not superior to placebo in terms of percent reduction in EASI Score from Baseline to Week 16; Test type: Superiority — Pairwise comparisons for each CBP-201 group vs placebo were performed and a serial gatekeeping procedure was used for multiplicity adjustment. Each CBP-201 group was compared with the placebo group in order from the highest dose (300 mg Q2W) to the lowest dose frequency (300 mg Q4W), until statistical significance at 0.05 level was not achieved; p = 0.0067, ANCOVA — Adjusted for multiplicity using a serial gatekeeping procedure at the 5% in descending order: 1. 300 mg dose Q2W 2. 150 mg Q2W 3. 300 mg Q4W vs placebo; The data were analyzed using an ANCOVA model with terms for treatment, baseline vIGA (moderate, severe), and baseline EASI; Mean Difference (Final Values) = 17.89, Standard Error of Mean 6.537
Statistical Analysis 3: Comparison: CBP-201 300 Q4W vs Placebo; The efficacy analysis includes comparing percentage reduction in EASI from baseline to Week 16 for CBP-201 300 mg Q4W regimen vs placebo. The sample size of the study was determined based on power calculations for the primary endpoint in patients receiving CBP-201 300 mg Q2W. Null hypothesis: CBP-201 300 Q4W is not superior to placebo in terms of percent reduction in EASI Score from Baseline to Week 16; Test type: Superiority — Pairwise comparisons for each CBP-201 group vs placebo were performed and a serial gatekeeping procedure was used for multiplicity adjustment. Each CBP-201 group was compared with placebo in order from highest dose (300 mg Q2W) to the lowest dose frequency (300 mg Q4W), until statistical significance at the 0.05 level was not achieved; p = 0.0004, ANCOVA — Adjusted for mulitplicity using a serial gatekeeping procedure at the 5% in descending order: 1. 300 mg dose Q2W 2. 150 mg Q2W 3. 300 mg Q4W vs placebo; The data were anlayzed using an ANCOVA model with terms for treatment, baseline vIGA (moderate, severe), and baseline EASI; Mean Difference (Final Values) = 23.83, Standard Error of Mean 6.575

2. Secondary Outcome: vIGA of 0/1 at Week 16
Description: Validated Investigator Global Assessment Score (vIGA) is assigned by the physician based on morphologic presentation of the disease in the clinic. The physician considers extent and severity of erythema, induration/papulation, lichenification, and oozing/crusting. A vIGA Score of 0=Clear, 1=Almost Clear, 2= Mild dermatitis, 3=Moderate dermatitis, and 4= Severe dermatitis. Patients are required to have a baseline IGA of 3 or 4. The response rate or percentage of patients achieving a vIGA of 0 or 1 (improved to clear or almost clear) at week 16 is the outcome.
Time Frame: Response Rate at 16 weeks
Population: All efficacy analyses were carried out using the FAS (all randomized subjects who received at least part of an SC dose of study drug), based on planned treatment assignment (ie, "as randomized").
Measure: Count of Participants; unit: Participants
Arm/Group | CBP-201 150 Q2W | CBP-201 300 Q2W | CBP-201 300 Q4W | Placebo
Number analyzed (Participants) | 57 | 57 | 56 | 56
Participants | 9 | 16 | 11 | 5
Statistical Analysis 1: Comparison: CBP-201 300 Q2W vs Placebo; Null hypothesis: CBP-201 300 Q2W is not superior to placebo in terms of the number of patients achieving a vIGA score of 0/1 (clear/almost clear) at Week 16; Test type: Superiority — The secondary efficacy analysis includes comparison of the number of patients achieving a vIGA score of 0/1 (clear/almost clear) at Week 16 for each CBP-201 300 mg Q2W vs placebo; p = 0.0089, Chi-squared — There were no adjustments for multiple comparisons. For IGA response, counts, percentage, and 95% CIs obtained using the Clopper-Pearson method and were presented for pairwise comparisons for each CBP-201 group vs. placebo; Difference in vIGA Response Rate = 28.1

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time the subject signed the informed consent and continued through the scheduled last visit (32 weeks after baseline visit), or if unresolved, until clinical recovery was complete.
Description: An adverse event (AE) is any untoward medical occurrence in a subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. All AEs will be reported along with causality (related or not related) and Severity (CTCAE grading 1-5). In addition, AEs will be considered AEs of Special Interest (AESI) if they are involve ophthalmic complications (conjunctivitis or keratitis). Serious AEs will be reported within 24 hours to the Sponsor and CRO.
Arm/Group | CBP-201 150 Q2W | CBP-201 300 Q2W | CBP-201 300 Q4W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57 | 1/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 1/57 | 0/57 | 2/56 | 2/56
Other Adverse Events (participants affected / at risk) | 26/57 | 21/57 | 34/56 | 31/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBP-201 150 Q2W (N=57) | CBP-201 300 Q2W (N=57) | CBP-201 300 Q4W (N=56) | Placebo (N=56)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBP-201 150 Q2W (N=57) | CBP-201 300 Q2W (N=57) | CBP-201 300 Q4W (N=56) | Placebo (N=56)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5) | 14 (14) | 8 (8)
COVID-19 (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 4 (4) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eye pruritis (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 1 (6) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT04444752/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT04444752/SAP_001.pdf
  • Informed Consent Form (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT04444752/ICF_002.pdf